CLINICAL TRIAL: NCT00377377
Title: Pharmacokinetics and Pharmacodynamic Effects of an Oral Ghrelin Agonist in Healthy Subjects
Brief Title: Oral Ghrelin Agonist in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKBB 67/04
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2006-07

CONDITIONS: Healthy Subjects
Keywords: GH release; Pharmacokinetics; Safety
MeSH Terms: interventions — macimorelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: EP1572 (ghrelin agonist) oral and duodenal application

SUMMARY:
EP01572 is a peptidomimetic growth hormone secretagogue, which has potent GH-releasing activity after intravenous administration.It is an analogue of the natural compound ghrelin. Since an oral delivery system would be preferable in many of the possible therapeutic indications, the pharmacological profile and the GH-releasing activity of increasing single, oral doses of EP01572 in healthy volunteers will be evaluated. In addition, the pharmacokinetics and pharmacological effects of EP01572 will be investigated after intraduodenal administration.

DETAILED DESCRIPTION:
EP01572 willbe given orally to 36 male subjects; the treatment will consist of one oral dose of either EP01572 or placebo (0.005, 0.05 and 0.5 mg/kg body weight). Subjects will receive one dose of EP01572 and placebo. Six subjects will receive two additional oral doses of EP01572: 0.125 and 0.25 mg/kg body weight. In another part, 6 subjects will receive the following treatments in a randomized order: 1) administration of a bolus of saline (placebo) to the small intestine; 2) intraduodenal (ID) administration of a bolus of EP01572 at 0.2 mg/kg body weight; 3) ID perfusion of a bolus of EP01572 at 0.35 mg/kg body weight; 4) ID perfusion of a bolus of EP01572 at 0.5 mg/kg body weight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males

Exclusion Criteria:

* Females

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42
Dates: Start 2005-11; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Growth hormone release
Pharmacokinetics

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, Principal Investigator — University Hospital, 4031 Basel Switzerland

REFERENCES:
- [Result] Piccoli F, Degen L, MacLean C, Peter S, Baselgia L, Larsen F, Beglinger C, Drewe J. Pharmacokinetics and pharmacodynamic effects of an oral ghrelin agonist in healthy subjects. J Clin Endocrinol Metab. 2007 May;92(5):1814-20. doi: 10.1210/jc.2006-2160. Epub 2007 Feb 6. PMID 17284637